CLINICAL TRIAL: NCT00427011
Title: A Multicenter, Open-Label Extension Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of E2007 In Patients With Parkinson's Disease Who Experience End-of-Dose "Wearing-Off" Motor Fluctuations
Brief Title: A Study of E2007 In Patients With Parkinson's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to lack of efficacy.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2007-A001-220
Record Dates: First submitted 2007-01-24; First posted 2007-01-26 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — perampanel

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E2007

INTERVENTIONS:
Drug: E2007 — E2007 2mg tablets. Dose (2mg, 4mg, 6mg or 8mg), is taken orally at nighttime.

SUMMARY:
Phase IIb open-label extension study for patients with Parkinson's Disease. All patients will receive active study drug. The study will involve outpatient visits only. Patients who completed Study E2007-A001-214 (Cohorts I and II) and who meet inclusion/exclusion criteria will be enrolled and enter the 12-week Titration Phase (from "Dispense Study Drug" at Week 0 [Visit 2] through Week 12 [Visit 7]) followed by the Maintenance Phase (from Week 12 [Visit 7] to end of study).

ELIGIBILITY:
INCLUSION CRITERIA

1. Male or female patients with idiopathic Parkinson's disease who have fulfilled the entry criteria for E2007-A001-214 and have completed that study up to and including the end of treatment (Day 70) visit and the Follow-up Visit at Day 91.

EXCLUSION CRITERIA

1. Pregnant or lactating women.
2. Women of child bearing potential unless infertile (including surgically sterile) or practicing effective contraception (e.g., intrauterine device or barrier method plus hormonal method). These patients must have a negative serum beta human chorionic gonadotropin (B-HCG) test at the initial visit (Visit 1) and urine pregnancy tests throughout the study. These patients must also be willing to remain on their current form of contraception for the duration of the study. Postmenopausal women may be recruited but must be amenorrhoeic for at least 1 year to be considered of nonchildbearing potential as determined by the investigator.
3. Patients who withdrew from Study 214 prior to the final efficacy visit for any reason, including lack of efficacy.
4. Patients with serious adverse events in Study 214 that are either ongoing or that are possibly or probably related to the study drug.
5. Patients with ongoing adverse events from Study 214 thought to be related to E2007.
6. Patients with a past (within the past 5 years) or present history of drug or alcohol abuse as per the criteria in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM IV).
7. Patients with a past (within 1 year) or present history of psychotic symptoms requiring antipsychotic treatment.
8. Patients with a past (within 1 year) or present history of suicidal ideation or suicide attempts.
9. Patients with active hepatic disease, significantly reduced hepatic function or significantly elevated liver enzymes (abnormal bilirubin or serum transaminase levels of more than 1.5 times the upper limit of the normal range).
10. Patients with clinically significant ECG abnormality, including prolonged QTc (defined as QTc >= 450 msec using Fridericia's correction).
11. Patients with clinically significant cardiovascular, metabolic, respiratory, renal, endocrinological, gastrointestinal diseases, psychiatric disorders, and bacterial or viral infections within the previous 30 days.
12. Patients who are currently taking medications known to induce the enzyme cytochrome P450 3A4.
13. Patients with current or prior treatment (within 4 weeks before entry visit) with tolcapone, methyldopa, budipine, reserpine, seroquel, or intermittent use of either liquid forms of levodopa or subcutaneous apomorphine.
14. Patients with previous stereotactic surgery (e.g., pallidotomy) for Parkinson's disease or with planned stereotactic surgery during the study period.
15. Patients receiving or with planned (next 6 months) deep brain stimulation.
16. Patients with conditions affecting the peripheral or central sensory system, unless related to Parkinson's disease (such as mild sensory or pain syndromes limited to OFF periods), that could interfere with the evaluation of any such symptoms caused by the study drug.
17. Patients with any condition that would make the patient, in the opinion of the investigator, unsuitable for the study.
18. Patients who have received an investigational product (other than E2007) within 4 weeks before screening.
19. Patients with clinically significant cognitive impairment (mini-mental state examination [MMSE] <24 or fulfilling DSM IV criteria for dementia due to Parkinson's disease).
20. Patients with any condition that could, in the opinion of the investigator, place the patient at increased risk or is likely to prevent completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Squillacote, MD, Study Director — Eisai Inc.
Locations (9):
- United States (9):
  - Pivotal Research Centers, Peoria, Arizona
  - Clinical Trials Incorporated, Little Rock, Arkansas
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Charlotte Neurological Services, Port Charlotte, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Agape Medical Research Center, Inc., Lubbock, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Perampanel: Subjects entered this open-label extension study from the double-blind core study E2007-A001-214 (NCT00165789), and included the placebo subjects. During the titration phase (lasting 12 weeks), subjects started on perampanel 2mg once daily for 2 weeks, 4 mg for 2 weeks, 6 mg for 2 weeks and finally, 8 mg until the end of the trial. Subjects remained on the same dose or had their dose reduced to their previously tolerated dose. Subjects were allowed to reduce the dose one or two steps, but only one step was allowed at a visit. Those subjects requiring more than two dose reductions were withdrawn. Subjects who did not tolerate the 2mg dose were discontinued from the study.
Period: Overall Study
Arm/Group | Perampanel
Started | 25
Completed | 0
Not Completed | 25
Not completed — Adverse Event | 10
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 2
Not completed — Other | 12

BASELINE CHARACTERISTICS:
Groups:
- Perampanel: Subjects entered this open-label extension study from the double-blind core study (E2007 A001 214), and included the placebo subjects. During the titration phase (lasting 12 weeks), subjects started on perampanel 2mg once daily for 2 weeks, 4 mg for 2 weeks, 6 mg for 2 weeks and finally, 8 mg until the end of the trial. Subjects remained on the same dose or had their dose reduced to their previously tolerated dose. Subjects were allowed to reduce the dose one or two steps, but only one step was allowed at a visit. Those subjects requiring more than two dose reductions were withdrawn. Subjects who did not tolerate the 2mg dose were discontinued from the study.
Arm/Group | Perampanel
Number analyzed (Participants) | 25
Age Continuous [Mean (Standard Deviation); unit: years] — Safety population.
  years | 69 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety population includes all subjects who received at least one dose of perampanel in this study.
  Participants
    Female | 7
    Male | 18
Race/Ethnicity, Customized [Number; unit: participants] — Race. Safety population.
  participants
    Caucasian | 23
    Black | 1
    Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline by Visit in Absolute OFF Time (Hours) During Open-label Extension Study
Description: OFF state is when medication has worn off and is no longer providing benefits with regard to stiffness, slowness, and tremor. This outcome measure was based on data collected through use of a patient diary.
Time Frame: Baseline, Week 12, Week 20, Week 32, Week 44, Week 56
Population: Safety population.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Perampanel (Placebo During Core Study); Perampanel (Perampanel During Core Study): Subjects entered this open-label extension study from the double-blind core study (E2007 A001 214), and included the placebo subjects. During the titration phase (lasting 12 weeks), subjects started on perampanel 2mg once daily for 2 weeks, 4 mg for 2 weeks, 6 mg for 2 weeks and finally, 8 mg until the end of the trial. Subjects remained on the same dose or had their dose reduced to their previously tolerated dose. Subjects were allowed to reduce the dose one or two steps, but only one step was allowed at a visit. Those subjects requiring more than two dose reductions were withdrawn. Subjects who did not tolerate the 2mg dose were discontinued from the study.
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel During Core Study)
Number analyzed (Participants) | 9 | 16
hours
  Week 12 (n=2,10) | -2.17 (4.714) | -1.18 (3.400)
  Week 20 (n=2,8) | -0.50 (4.714) | -0.29 (3.261)
  Week 32 (n=2,10) | -0.25 (6.718) | -0.97 (2.765)
  Week 44 (n=0,7) | NA (NA) — Insufficient data due to early withdrawals/study termination. | -0.81 (2.678)
  Week 56 (n=0,0) | NA (NA) — Insufficient data due to early withdrawals/study termination. | NA (NA) — Insufficient data due to early withdrawals/study termination.

2. Secondary Outcome: Mean Change From Baseline by Visit in Absolute ON Time (Without Dyskinesias or With Nontroublesome Dyskinesias) (Hours) During Open-label Extension Study
Description: ON state is when medication is providing benefits with regard to stiffness, slowness, and tremor. This outcome measure was based on data collected through use of a patient diary.
Time Frame: Baseline, Week 12, Week 20, Week 32, Week 44, Week 56
Population: Safety population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel During Core Study)
Number analyzed (Participants) | 9 | 16
hours
  Week 12 (n=2,10) | 1.42 (3.889) | 1.15 (3.162)
  Week 20 (n=2,8) | -0.17 (2.357) | 0.69 (1.838)
  Week 32 (n=2,10) | 0.08 (3.418) | 1.18 (2.905)
  Week 44 (n=0,7) | NA (NA) — Insufficient data due to early withdrawals/study termination. | 0.93 (2.757)
  Week 56 (n=0,0) | NA (NA) — Insufficient data due to early withdrawals/study termination. | NA (NA) — Insufficient data due to early withdrawals/study termination.

3. Secondary Outcome: Mean Change From Baseline by Visit in UPDRS Part II (ADL) in OFF State (Hours) During Open-label Extension Study
Description: Unified Parkinson's Disease (PD) Rating Scale (UPDRS) is a standardized assessment of the symptoms and signs of PD. Part II assesses Activities of Daily Living (ADL) based on 13 items, such as speech, hygiene, and falling. Participants receive a score of 0-4 points per item, with a higher score indicating more severe symptoms. Range of possible total scores, 0 to 52. ON state is when medication is providing benefits to mobility, slowness, and stiffness. OFF state is when medication has worn off and is no longer providing benefits with regard to stiffness, slowness, and tremor.
Time Frame: Baseline, Week 12, Week 20, Week 32, Week 44, Week 56
Population: Safety population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel During Core Study)
Number analyzed (Participants) | 9 | 16
scores on a scale
  Week 12 (n=2,11) | 7.50 (0.707) | -1.27 (4.777)
  Week 20 (n=1,12) | 8.00 (NA) — Insufficient data due to early withdrawals/study termination. | -1.33 (4.979)
  Week 32 (n=1,11) | NA (NA) — Insufficient data due to early withdrawals/study termination. | 0.55 (5.007)
  Week 44 (n=1,8) | 2.00 (NA) — Insufficient data due to early withdrawals/study termination. | 1.63 (5.706)
  Week 56 (n=0,5) | NA (NA) — Insufficient data due to early withdrawals/study termination. | 1 (8)

4. Secondary Outcome: Mean Change From Baseline by Visit in UPDRS Part III (Motor) Score in ON State (Hours) During Open- Label Extension Study
Description: The UPDRS is a standardized assessment of the symptoms and signs of Parkinson's Disease. Part III assesses motor activity, based on 14 items, such as gait, facial expression, and rigidity. Participants receive a score of 0-4 points per item, with a higher score indicating more severe symptoms. Range of possible total scores, 0 to 56. ON state is when medication is providing benefits with regard to stiffness, slowness, and tremor.
Time Frame: Baseline, Week 12, Week 20, Week 32, Week 44, Week 56
Population: Safety population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel During Core Study)
Number analyzed (Participants) | 9 | 16
scores on a scale
  Week 12 (n=3,12) | -3.67 (3.055) | -2.67 (3.627)
  Week 20 (n=2,12) | -1.00 (7.071) | -3.25 (8.996)
  Week 32 (n=2,11) | -8.00 (2.828) | -1.91 (6.395)
  Week 44 (n=2,8) | -5.50 (7.778) | -3.63 (8.210)
  Week 56 (n=0,5) | NA (NA) — Insufficient data due to early withdrawals/study termination. | -6.40 (7.829)

ADVERSE EVENTS:
Arm/Group | Perampanel
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (N=25)
Dysarthria (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Confusional State (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (N=25)
Cataract (Eye disorders) | 2
Vision Blurred (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Gait Disturbance (General disorders) | 2
Irritability (General disorders) | 2
Oedema Peripheral (General disorders) | 3
Excoriation (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 3
Skin Laceration (Injury, poisoning and procedural complications) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Balance Disorder (Nervous system disorders) | 3
Coordination Abnormal (Nervous system disorders) | 4
Disturbance in Attention (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 8
Dyskinesia (Nervous system disorders) | 6
Hyporeflexia (Nervous system disorders) | 2
ON and OFF Phenomenon (Nervous system disorders) | 8
Somnolence (Nervous system disorders) | 7
Tremor (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 2
Confusional State (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 2
Urinary Incontinence (Renal and urinary disorders) | 3
Orthostatic Hypotension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Due to early termination, a limited number of subjects (n=26) were screened for inclusion in the study and only 25 subjects were analyzed. The majority of subjects did not reach the scheduled Week 56 assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No